CLINICAL TRIAL: NCT05518890
Title: Effect of Short-term Negative Energy Balance With or Without Exercise on Systemic Biomarkers in Patients With Knee Osteoarthritis
Brief Title: Effect of Energy Restriction and Exercise for Knee Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Bath (Other)
Collaborators: University of Oxford (Other)
Responsible Party: Principal Investigator, James Bilzon, Professor James Bilzon, University of Bath
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20/SW/0063
Record Dates: First submitted 2022-03-29; First posted 2022-08-29 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Diet; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diet Only (Experimental): Reduced calorie intake by 5000kcals per week over a 4 week period
  Interventions: Other: Diet Only
- Diet plus Exercise (Experimental): Reduced calorie intake by 5000kcals per week over 4 weeks with the addition of five 30 minute exercise sessions per week on a cycle ergometer. The exercise in intensity will be progressive and perceptually based and monitored by the investigators.
  Interventions: Other: Diet plus Exercise

INTERVENTIONS:
Other: Diet Only — Participants caloric intake will be reduced by 5000kcal per week over 4 weeks
  Arms: Diet Only
Other: Diet plus Exercise — Participants caloric intake will be reduced by 5000kcal per week over 4 weeks. Participants will also be asked to perform 5x30 minute cycling exercise sessions at home. Each week the intensity of exercise will be increased (week 1 = RPE 12, week 2 = RPE 13, week 3 = RPE 14, week 4 = RPE 15)
  Arms: Diet plus Exercise

SUMMARY:
The investigators are looking at the effects of energy restriction, with or without exercise on markers of inflammation in individuals with knee osteoarthritis. There will be a 4 week 'wash-in' period where participants will maintain their normal lifestyle, followed by a 4 week 'intervention period' where participants will be randomised into either the diet alone group or the diet plus exercise group.

DETAILED DESCRIPTION:
Knee Osteoarthritis is a condition that causes pain, reduced physical function and quality of life. Long-term studies have shown that exercise and substantial weight loss can cause improvements in these factors. Individuals with knee Osteoarthritis might have changes in their joint that can be seen with x-ray images. However, this is not guaranteed, and imaging does not always detect changes that occur with interventions that cause improved symptoms. As a result, there is interest in biological markers (biomarkers) as another way of monitoring Osteoarthritis. These markers can be examined in biological tissues, with samples measured in blood easier to obtain than those taken from the fluid within the joint itself. Historically, Osteoarthritis was thought of as a disease caused by mechanical factors but we are now aware that inflammation also plays a part.

Therefore, the investigators aim to test a short -term diet/exercise intervention that has been show to improve inflammation in other populations, in individuals with knee osteoarthritis. Importantly, this will allow the investigators to see if reducing food intake alone or doing this with regular exercise can improve outcomes without substantial weight loss. The investigators will ask individuals to participate in one of two groups where they will first be asked to continue their normal lifestyle for 4 weeks to check the stability of outcomes. The investigators will then ask individuals to either reduce their food intake by 5000 calories per week, or do this while also completing moderate intensity cycling exercise 5 times a week for 4 weeks. At the start and end of each period the investigators will collect a blood sample to assess markers of inflammation and disease related processes. The investigators will also conduct questionnaire measurements, tests of physical function and experimental pain and scan participants to establish body composition.

ELIGIBILITY:
Inclusion Criteria:

* Male or post-menopausal females
* Clinically diagnosed with knee Osteoarthritis including radiographic confirmation
* Oxford Knee Score ≥20 to ≤35 for index knee
* Aged 45-69 years
* BMI ≥27.5kg/m2 to ≤40.0 kg/m2
* Daily physical activity level <2.00

Exclusion Criteria:

* Inability to undertake cycling exercise safely
* Use of prescribed anti-inflammatory medication
* Current smoker (or having quit <6months ago)
* Has a diagnosis of diabetes or other metabolic disorder
* Use of other medications that might interfere with study outcomes
* Recent (within last 3 months) change in body mass of >5%
* Currently engaged in an ongoing programme of physiotherapy treatment
* Currently on waiting list or having had surgery for Osteoarthritis on the index knee (prior OA related surgery permitted on other knee as long as this is greater than 12 months prior to enrolment)
* Having had major hip/knee surgery within preceding 12 months
* Individuals with a blood pressure of greater than 180/110
* Currently pregnant or intending to become pregnant during the study

Ages: 45 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in hsCRP | 0, 4 and 8 weeks
  Measured in mg/L via immunoassay

SECONDARY OUTCOMES:
Other Systemic Biomarkers | 0, 4 and 8 weeks
  Measured in pg/ml via electrochemiluminescence
  * Interleukin-1 Beta
  * Interleukin-1Receptor Antagonist
  * Interleukin- 4
  * Interleukin- 6
  * Interleukin- 8
  * Interleukin- 10
  * Interleukin- 13
  * Interleukin-17A
  * Interleukin-18
  * Tumor Necrosis Factor- alpha
The Knee Injury and Osteoarthritis Outcome Score (KOOS) | 0, 4 and 8 weeks
  Pain, Symptoms, Activity of daily living, Sport/Rec, Quality of Life subscales. Each subscale has a minimum score of 0% and a maximum score of 100%, with lower values representing worse outcomes.
EQ-5D-5L Health Questionnaire | 0, 4 and 8 weeks
  Mobility, Self-care, Usual activities, Pain/discomfort and Anxiety/depression. Each of the five dimensions comprising the EQ-5D descriptive system is divided into five levels of perceived problems:
  LEVEL 1: indicating no problem LEVEL 2: indicating slight problems LEVEL 3: indicating moderate problems LEVEL 4: indicating severe problems LEVEL 5: indicating unable to/extreme problems
  A unique health state is defined by combining one level from each of the five dimensions.
SF-36 Questionnaire | 0, 4 and 8 weeks
  Physical functioning, Bodily pain, Role limitations due to physical health problems, Role limitations due to personal or emotional problems, Emotional well-being, Social functioning, Energy/fatigue, and General health perceptions. Scores for each domain range from 0 to 100, with a higher score defining a more favourable health state.
Visual Analogue Scale (VAS) Pain | 0, 4 and 8 weeks
  0-10 scale Higher scores indicate worse pain
30-second chair stand test | 0, 4 and 8 weeks
  Repetitions
40m fast paced walk | 0, 4 and 8 weeks
  meters/second
Stair climb | 0, 4 and 8 weeks
  seconds
Timed up and go test | 0, 4 and 8 weeks
  seconds
Mechanical Detection Threshold | 0, 4 and 8 weeks
  millinewtons (mN)
Pressure Pain Threshold | 0, 4 and 8 weeks
  Newtons (N)
Body Mass Index | 0, 4 and 8 weeks
  kg/m2
Hip and Waist Circumference | 0, 4 and 8 weeks
  centimetres
Body Composition | 0, 4 and 8 weeks
  Change in body composition via Dual Energy XX-Ray Absorptiometry scan
Markers of metabolic health | 0, 4 and 8 weeks
  mmol/L
  * Glucose
  * Non-Esterified Fatty Acids
  * Triglycerides
  * Total cholesterol
  * Low Density Lipoprotein Cholesterol
  * High Density Lipoprotein Cholesterol

CONTACTS AND LOCATIONS:
Overall Officials: James Bilzon, PhD, Principal Investigator — University of Bath
Locations (1):
- University of Bath, Bath, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Anonymous individual data for all outcomes may be made available.

DOCUMENTS (2):
  • Study Protocol (2020-10-13): https://cdn.clinicaltrials.gov/large-docs/90/NCT05518890/Prot_000.pdf
  • Informed Consent Form (2021-01-14): https://cdn.clinicaltrials.gov/large-docs/90/NCT05518890/ICF_001.pdf